CLINICAL TRIAL: NCT01152034
Title: Effect of Psychoeducational Group Therapy Model for Bipolar Disorder Patients
Brief Title: MAPS Group Therapy Model for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chen-Ju Lin, senior visiting staff, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMH-I-S-662
Record Dates: First submitted 2010-06-22; First posted 2010-06-29 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Bipolar Disorder; Suicide
Keywords: Bipolar disorder; psychosocial intervention; group therapy; relapse prevention; parasuicide; Recurrence; hospitalization; Medication adherence; Self-Injurious Behavior; Quality of Life
MeSH Terms: conditions — Bipolar Disorder; Suicide; Suicide, Attempted; Recurrence; Medication Adherence; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychoeducation group therapy (Experimental): The structured group program comprised of an initial block of 12 weekly sessions with three additional monthly booster sessions, designed to support participants in the application of knowledge and skills to everyday life situations. All participants also received standard psychiatric care as well.
  Interventions: Behavioral: psychoeducation group therapy
- Treat as Usual (Placebo Comparator): Patients who were assigned to the control group received standard psychiatric care and standard pharmacological treatment without group-based psychosocial intervention. Weekly phone calls to the control group over the initial 12 weeks were controlled for any extra contact time with researchers outside of the structured intervention group.

INTERVENTIONS:
Behavioral: psychoeducation group therapy — This program consists of 15 sessions of closed group, with each session lasting 120 minutes, each aims at improving four main issues: illness awareness, early detection of prodromal symptoms and recurrences, treatment adherence, and lifestyle regularity. The program will be in groups of 6-12, conducted by two experienced therapists. The structure of each session consists of 30-40 minutes talk on the topic of the day, followed by an exercise related to the issue and a discussion.
  Arms: Psychoeducation group therapy

SUMMARY:
This study aims to develop the MAPS(M,Monitoring;A,Assessing;P,Preventing or Reducing Relapse;S,Smart goal setting) group therapy model for bipolar disorder patients as other adjuvant clinical treatment and develop the instruments for evaluating the severity of bipolar symptoms. The investigators insist to provide the psychosocial intervention for bipolar patients in the general hospital and offer appropriative adjuvant intervention except current psychiatric biological treatment.

This study is a one-year project. First, the investigators like to translate the Depression, Anxiety and Stress Scale (DASS) and the Altman Self-Rating Scale for Mania (ASRM) to Chinese and finish the reliability and validity study. Second, the investigators would like to develop the MAPS group therapy to enhance bipolar patients' insight, increased life quality and decrease suicidal ideation. This study is a case control study. All cases recruit from the psychiatric outpatient department of one medical center. The inclusion criteria are diagnosed as bipolar disorder, age from 18 to 65 and agree to sign the inform consent. The excluded criteria are hard to communicate, with acute psychiatric feature and severe physical illness. The investigators plan to hold the MAPS group three times and predetermine to recruit totally 30 patients as the case group. As to the control group, the investigators also recruit from the psychiatric outpatient department and those who treat as usual by control their gender, age and the same diagnosis as bipolar disorder. The only one different factor between the case group and the control group was attending the MAPS group therapy or not. In MAPS group therapy, two facilitators work with ten clients with twelve weekly sessions and three monthly booster sessions. Self-report rating scales (DASS and ASRM) are completed at the beginning of each session. The investigators use DASS and ASRM to evaluate the severity of bipolar symptoms; BSS for suicidal ideation; SF-36 for life quality. The hypothesis is "patients attended to MAPS group therapy have better symptoms control, lower suicidal ideation, better life quality and less use emergency department or admissions than those who didn't attend the group therapy".

ELIGIBILITY:
Inclusion Criteria:

* bipolar disorder outpatients in remission, defined as Young Mania Rating Scale score < 6, Hamiltone Depression Rating Scale-17 < 8
* age 18 to 65 years old
* speaking Mandarin
* agree to sign the inform consent

Exclusion Criteria:

* Those who were hard to communicate such as mental retardation, hearing impairment and etc
* with acute psychotic feature
* with severe physical illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The main outcome measures are time to recurrence a new acute bipolar episode | every 3 months for up to 12 months after enrollment
  This is defined as the time (days) elapsed between baseline and the emergence of a new acute episode according to DSM-IV criteria and scores above or equal to 20 on the YMRS for manic recurrence; above or equal to 12 for hypomanic recurrence; above or equal to 17 on the HRSD-17 for depressive recurrence; and above or equal to 20 on the YMRS and 12 on the HRSD-17 for mixed recurrence.

SECONDARY OUTCOMES:
Number of recurrences | every 3 months for up to 12 months after enrollment
  The number of recurrences, separating for type of episode (manic, hypomanic, mixed or depressive) will also be recorded as a secondary outcome measure.
Time spent ill | every 3 months for up to 12 months after enrollment
  Another secondary outcome measure is time spent ill. The investigators obtain this data by prospectively registering the number of days that a participant fulfilled criteria for a specific episode.
Psychiatric outpatient adherence and drug compliance | every 3 months for up to 12 months after enrollment
  The medication compliance questionnaire reported compliance with any prescribed mood stablizers.(Lam DH, et al. 2000, 2005) Respondents had a choice of noting whether the patient in the past month had (1) never missed taking their medication, (2) missed taking it once or twice, (3) missed taking it between three to seven times, (4) missed taking it more than seven times, or (5) stopped taking it altogether.
Numbers and time of emergency use and hospitalization | every 3 months for up to 12 months after enrollment
  The number of hospitalizations, reasons for admission and total number of days that the participant remained hospitalized will also be recorded during follow-up period.
Suicidal ideation and number of suicidal attempt | every 3 months for up to 12 months after enrollment
  The Chinese version of Scale for Suicide Ideation had been translated and the excellent psychometric properties for measuring suicidal ideation in Chinese populations were done (Zhang and Brown, 2007). The BSS and the suicidal attempts will be re-assessed every 3 months or whenever a new episode was suspected by the psychiatrist in charge of the participant.
The life quality of bipolar patients | every 3 months for up to 12 months after enrollment
  This SF-36 Taiwan standard version was developed in 1996 following the protocol by the International Quality of Life Assessment (IQOLA) Project. The protocol includes forward and backward translation, focus group discussion, pilot testing, and extensive psychometric analysis of the translation. (Fuh JL et al, 2000; Chang DF,et al, 2000).The SF-36 Taiwan standard version will be also repeated every 3 months or whenever a new episode was suspected by the psychiatrist in charge of the participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan